CLINICAL TRIAL: NCT01115660
Title: AVAIL interVention Trial (Adherence Evaluation After Ischemic Stroke - Longitudinal): Pilot Protocol
Brief Title: Stroke Education Intervention Trial - Pilot
Acronym: AVAIL II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00019690; 5U18HS016964 (AHRQ)
Record Dates: First submitted 2010-05-02; First posted 2010-05-04 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-12

CONDITIONS: Ischemic Stroke; Intracranial Hemorrhage; Transient Ischemic Attack
Keywords: stroke; patient education; medication adherence
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages; Ischemic Attack, Transient; Stroke; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stroke education (Experimental): Patients in this arm receive a telephone call by a medication coach who reviews their condition and importance of adherence to medication regimen.
  Interventions: Behavioral: stroke education
- control arm (No Intervention): Subjects in this arm received instruction at hospital discharge and a 3-month follow-up call to collect study data.

INTERVENTIONS:
Behavioral: stroke education — call by medication coach 2 weeks after hospital discharge
  Arms: stroke education

SUMMARY:
The objectives of the trial of a medication-coach program for patients with stroke or transient ischemic attack are to pilot test the study design, the intervention components and the data collection forms and refine them for a larger trial whose goal will be to improve long-term adherence to stroke prevention medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Wake Forest University Baptist Medical Center (WFUBMC) over age 18
* Diagnosed with acute ischemic stroke, transient ischemic attack or intracranial hemorrhage
* provide consent to participate

Exclusion Criteria:

* discharged to nursing home, acute rehabilitation center, inpatient hospice, or other acute hospital
* homeless
* non-English speakers
* patient and proxy unable to participate in telephone conversation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Peterson, MD, MPH, Principal Investigator — DCRI
Locations (1):
- WFUBMC, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Sides EG, Zimmer LO, Wilson L, Pan W, Olson DM, Peterson ED, Bushnell C. Medication coaching program for patients with minor stroke or TIA: a pilot study. BMC Public Health. 2012 Jul 25;12:549. doi: 10.1186/1471-2458-12-549. PMID 22830539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled patients in 2010 at Wake Forest Baptist Medical Center
Pre-assignment Details: Patients assigned to intervention arm and control arm, consecutively.
Groups:
- Control Arm: Patients received standard discharge counseling but no 2-week follow-up call.
Period: Overall Study
Arm/Group | Stroke Education | Control Arm
Started | 20 | 10
Completed | 19 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke Education | Control Arm | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Median Age | 61 (7) [55 to 70] | 59 (10) [47 to 67] | 61 (8) [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention (Ability to Reach Patients at 3 Months)
Description: Number of patients contacted at 3 months
Time Frame: 3 months
Population: All eligible patients who also were available at 3 months for post-intervention follow-up call.
Measure: Number; unit: number of patients contacted
Groups:
- Control: standard of care
Arm/Group | Stroke Education | Control
Number analyzed (Participants) | 19 | 10
number of patients contacted | 16 | 10

2. Secondary Outcome: Follow up Appointment With MD
Description: Follow up appointment with primary care provider since stroke
Time Frame: 3 months
Population: Patients who were contacted at 3 months
Measure: Number; unit: participants
Arm/Group | Stroke Education | Control
Number analyzed (Participants) | 16 | 10
participants | 15 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Arm/Group | Stroke Education | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Adverse events not collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No